CLINICAL TRIAL: NCT02571647
Title: Evaluation of Screening for Visual Disorders of the Old Subject in Consultation Memory
Acronym: EVAM
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0219
Record Dates: First submitted 2015-10-05; First posted 2015-10-08 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Visual Disorders
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non interventional study — Patients agreeing to participate in the study will have a cognitive assessment and geriatric assessment, carried out according to usual practices and grids clinical gerontology cluster.
  They will benefit in addition to a noninvasive screening and risk-free ophthalmic (visual acuity, intraocular pressure, examination of the eyelids and fundus).

SUMMARY:
Visual disorders are often overlooked in the treatment of cognitive disorders of the elderly. Yet the visual deficit impacts the quality of life, the evolution of the autonomy and psycho-behavioral disorders in cognitive diseases. The main objective of the study is to evaluate the prevalence of visual disorders among elderly patients at consultant outpatient center of Nantes clinical gerontology as part of the consultation geriatric memory. Secondary objectives are to describe ophthalmological diseases detected and taken into the proposed ophthalmic load, to determine if there are associations between eye diseases and cognitive disorders, to estimate the proportion of patients who may have an ophthalmologic evaluation to determine the cognitive profiles and geriatric evaluation and ocular pathological, depending on the assessment of arterial stiffness. The results of this study will build a testing strategy to promote access of older patients with cognitive impairment to vision care.

ELIGIBILITY:
Inclusion Criteria:

* Elderly over 65 years,
* Subject to consultation from memory Clinical Gerontology ambulatory center Nantes University Hospital
* Current use of spoken French
* Patient (or legal guardian, if applicable) has given its written consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Life expectancy lower 1 year
* Mobility limitation preventing the installation retinal
* Major disorders and productive behavior does not allow participation in diagnostic procedures.
* Inability to respond to instructions when performing ophthalmological examinations.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients eligible for the study will be all patients 65 and older, in consultation from memory or day hospital Clinical Gerontology ambulatory center at Nantes University Hospital.
  Geriatrician who will see the patient Clinical Gerontology ambulatory center be informed of the study and gather written consent and that of his legal representative, if applicable.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with presence of an ophthalmological disease (symptomatic or not) after clinical evaluation. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Gilles BERRUT, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France